CLINICAL TRIAL: NCT01494298
Title: Preliminary Analysis of Lipoprotein Subclasses, Apoprotein Levels, and Genetic Architecture of African-American Males With Type 2 Diabetes. Lipids in African Americans With Type 2 Diabetes
Brief Title: Study of Cholesterol Levels and Types in African Americans With Type 2 Diabetes
Acronym: LAAD
Status: Completed | Type: Observational
Sponsor: Mercer University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Emory University (Other); Celera Genomics (Industry)
Responsible Party: Principal Investigator, Gina J. Ryan, Clinical Associate Professor, Mercer University
Other Study IDs: H1105110
Record Dates: First submitted 2011-12-15; First posted 2011-12-16 (Estimated); Results first posted 2013-12-13 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-10

CONDITIONS: Type 2 Diabetes; African American; Cholesterol; Lipoprotein; Apolipoprotein
Keywords: Type 2 diabetes; African American; cholesterol; lipoprotein; apolipoprotein
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We will retain a sample of serum, plasma and whole blood.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- T2DM: African-American men with type 2 diabetes who are not taking cholesterol-lowering medications.
- Control: African-American men without type 2 diabetes who are not taking cholesterol-lowering medications.

SUMMARY:
Compared to other races, African-Americans with type 2 diabetes have different cholesterol levels, specifically triglycerides and low density lipoprotein. Recent data has shown the not only are cholesterol levels important in determining the risk for cardiovascular disease, but the size of the cholesterol particles and surface proteins on the cholesterol particles are also important. The objective of this study is to determine if African-American males with diabetes have different particle size, surface proteins, and cholesterol genetic links than African-American male without diabetes and Caucasian-American males with and without diabetes.

African-American males with type 2 diabetes and not taking lipid-lowering medications are the current target population.

After obtaining an informed consent, a complete medical history will be obtained and subjects will be examined, noninvasively, for physical signs of elevated cholesterol levels. Afterwards, blood samples [one venous puncture, 6 tubes (21 mL total)] will be obtained. Blood samples will be coded, sent to Berkeley Heart Lab and/or Clinical Laboratory Services, and undergo genetic testing at Mercer University College of Pharmacy and Health Sciences.

Confidentiality of the subjects will be explained in the consenting process to the subjects. All subject samples and information will be coded. Each subject will be given a subject number upon consenting and this will be used throughout the study. All pertinent information of the subjects will be listed under the designated number, but will not be associated with that patient.

ELIGIBILITY:
Inclusion Criteria:

* Male
* African American by self-report
* Subjects will be defined as having diabetes if they are diagnosed with diabetes per the American Diabetes Association guidelines
* Subjects without diabetes or impaired glucose tolerance will have a fasting blood glucose <100 mg/dL and/or glycosylated hemoglobin(A1C) <6.5%.

Exclusion Criteria:

* Females
* Self report of race or ethnicity other than African
* Currently taking any lipid-lowering medications

Ages: 18 Years to 79 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a cross-sectional epidemiologic study in which the lipoprotein subclasses, apolipoprotein levels, and genetic polymorphisms of African-American men with type 2 diabetes will be compared to African-American men without diabetes.
Sampling Method: Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2011-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Grady Health System, Atlanta, Georgia
  - Mercer Univeristy College of Pharmacy and Health Sciences, Atlanta, Georgia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Inclusion criteria were male gender, African American by self report and not taking of lipid-lowering medications. Subjects with diabetes were recruited from the Grady Diabetes Clinic in Atlanta, Georgia. Control subjects were recruited from the general Metro-Atlanta Area and had to have a fasting blood glucose <100 mg/dL.
Pre-assignment Details: 1 subject was excluded from the diabetes group because he had type 1 diabetes
  Exclusion from control group 1- was taking lipid lowering medications
  1 - was not possible to do venous blood draw 5 - FBG between 100-126 mg/dL 2 - FBG>126 and were reassigned to diabetes group
Groups:
- T2DM: African American men with type 2 diabetes and not taking cholesterol-lowering medications.
- Controls: African American men without type 2 diabetes and not taking cholesterol-lowering medications.
Period: Overall Study
Arm/Group | T2DM | Controls
Started | 56 | 55
Completed | 54 | 47
Not Completed | 2 | 8
Not completed — Protocol Violation | 2 | 8

BASELINE CHARACTERISTICS:
Population: The primary objective of this project was to determine the difference in Apo B levels in African-American men with and without diabetes.To achieve a power of 80%, 48 subjects in each group were needed to detect 15 mg/dL difference in ApoB levels, assuming a standard deviation of 26 mg/dL if alpha was set at 0.05.
Groups:
- T2DM: African American Men with Type 2 Diabetes
- Controls: African American Men without diabetes
- Total: Total of all reporting groups
Arm/Group | T2DM | Controls | Total
Number analyzed (Participants) | 54 | 47 | 101
Age Continuous [Mean (Standard Deviation); unit: Years] | 52 (8) | 44.5 (13.1) | 48.5 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 54 | 47 | 101
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 54 | 47 | 101
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 54 | 47 | 101

OUTCOME MEASURES:

1. Primary Outcome: ApoB Levels in African American Men With Diabetes and Those Without.
Description: Apolipoprotein B Age adjusted least square means are reported because of baseline differences in ages.
Time Frame: At study entry
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | T2DM | Controls
Number analyzed (Participants) | 54 | 47
mg/dL | 80 (3) | 65 (3)
Statistical Analysis 1: Comparison: T2DM vs Controls; Hypothesis - There will be differences in ApoB between AA with T2DM and those without. To achieve a power of 80%, 48 subjects in each group were needed to detect 15 mg/dL difference in ApoB levels, assuming a standard deviation of 26 mg/dL if alpha was set at 0.05. Continuous data were compared using a Students t-test and categorical data were compared using test; Test type: Superiority or Other; p = 0.002, t-test, 2 sided — The control group average age was 6 years lower(P=0.001). Results were adjusted via a logistic regression and presented as age-adjusted means and SE. The unadjusted differences had similar results

2. Secondary Outcome: LDL Density in African American Males With Diabetes and Those Without Diabetes
Description: LDL size subclassification was divided into the following groups (from largest size to smallest size): LDL I, LDL IIa, LDL IIb, LDL IIIa, LDL IIIb, LDL IVa, LDL IVa, and LDL IVb.
  For differences posted P<0.05 for LDL I, LDL IIb, LDL IIIa, and LDL IIIa +b
Time Frame: at entry
Measure: Least Squares Mean (Standard Error); unit: percentage of total LDL particles
Groups:
- T2DM: African-American men with type 2 diabetes who are not taking cholesterol lowering medications
- Controls: African-American men without type 2 diabetes who are not taking cholesterol lowering medications
Arm/Group | T2DM | Controls
Number analyzed (Participants) | 54 | 47
percentage of total LDL particles
  LDL I | 21 (1) | 29 (1)
  LDL IIa | 24 (1) | 27 (1)
  LDL IIb | 29 (1) | 24 (1)
  LDL IIIa | 18 (1) | 13 (1)
  LDL IIIb | 3.3 (0.3) | 3.4 (0.3)
  LDL IVa | 2.8 (0.2) | 2.8 (0.2)
  LDL IVb | 1.4 (0.1) | 1.3 (0.1)
  LDL IIIa +b | 21 (2) | 16 (2)

3. Secondary Outcome: Lipoprotein a [Lp(a)] in African Americans With Diabetes and Without.
Time Frame: at study entry
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | T2DM | Controls
Number analyzed (Participants) | 54 | 47
mg/dL | 43 (5) | 45 (5)
Statistical Analysis 1: Comparison: T2DM vs Controls; Test type: Superiority or Other; p = 0.84, t-test, 2 sided

ADVERSE EVENTS:
Description: Since this was an observational study, serious and/or other non-serious adverse events were not collected/assessed.
Arm/Group | T2DM | Controls
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less